CLINICAL TRIAL: NCT05573620
Title: Training University Students Through Acceptance and Virtual Reality for Coping Public Speaking Fear: a Clinical Trial
Brief Title: ACT and Virtual Reality for Public Speaking Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIPI/19/052
Record Dates: First submitted 2022-09-13; First posted 2022-10-10 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Public Speaking Fear
MeSH Terms: conditions — Glossophobia

STUDY DESIGN:
Intervention Model Description: Randomization assigned participants to 3 arms:
  * in vivo exposure
  * virtual reality
  * waiting list
Who Masked: Participant
Masking Description: Participants did not know that two different treatments were delivered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ACT+In vivo exposure (Experimental): 5 individual weekly sessions which included ACT methods + in vivo exposure
  Interventions: Behavioral: ACT; Behavioral: In vivo exposure:
- ACT+Virtual reality (Experimental): 5 individual weekly sessions which included ACT methods + virtual reality
  Interventions: Behavioral: ACT; Behavioral: Virtual Reality
- Waiting list (No Intervention): Participants assigned to Waiting List arm waited for 5 weeks before receiving treatment (i.e., after completing the measures they continued in the study and then were randomly assigned to ACT+in vivo exposure or ACT+virtual reality arms).

INTERVENTIONS:
Behavioral: ACT — Acceptance and Commitment Therapy methods were focused on promoting Values clarification, Acceptance, Cognitive defusion, Committed action and Flexible attention to the present moment, and included 'The dreamed professional exercise' -variation on '"imagine your funeral" exercise'-, Ship's captain metaphor, Imaginal exposure, Physicalizing exercise, and Watching thoughts as graffiti.
  Arms: ACT+In vivo exposure; ACT+Virtual reality
Behavioral: In vivo exposure: — The audience was made up of university students. Every session included a 12 minute oral presentation. Participants were asked to improvise a talk about a new topic (e.g. violence against women, education system in Spain…). Participants had 3 minutes to prepare their speech. Difficulty increased based on each participant's pre assessment (topics and distractors as ringtones, audience whispering...)
  Arms: ACT+In vivo exposure
Behavioral: Virtual Reality — Virtual reality was delivered through Psious platform distributed in Spain by TEA and through a Virtual Reality equipment that included a Samsung S7 mobile and Samsung Gear VR glasses.
  Every session included a 12 minute oral presentation. Participants were asked to improvise a talk about a new topic (e.g. violence against women, education system in Spain…). Participants had 3 minutes to prepare their speech. Difficulty increased based on each participant's pre assessment (topics and distractors as ringtones, audience whispering...)
  Arms: ACT+Virtual reality

SUMMARY:
Investigation of Acceptance and Commitment Therapy (ACT) for the psychological treatment of public speaking fear. Two ACT-based treatment delivery modalities (in vivo exposure vs. virtual reality) were compared.

DETAILED DESCRIPTION:
After being informed about the study, all patients giving written informed consent will be assessed to determine eligibility for study entry.

The clinical trial will include a control group (waiting list).

Patients who meet eligibility requirements will be assigned to a waiting list, in vivo exposure and Virtual Reality.

Psychological intervention consisted in a 5-session individual face-to-face delivered ACT-based treatment.

The participants will be assessed through self-report instruments and observational measurements before and after treatment and at 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Student at European University of Madrid, Spain
* Significant social anxiety (LSAS Liebowitz Social Anxiety Scale)
* Subjective fear intensity and interference > 5/10

Exclusion Criteria:

* Alcohol or drugs abuse
* Psychotropic drug consume
* Following psychological/psychiatric treatment
* Serious mental disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Public Speaking Self-confidence questionnaire PRCS (Paul, 1966) | Change from Baseline psychological inflexibilty at 4 months
  'Public Speaking Self-confidence questionnaire' assesses public speaking fear. It is a 12-item, five-point Likert-type scale. Scores range between 12 and 60. Higher the score in the questionnaire, indicate higher levels of public speaking fear and worse outcome.

SECONDARY OUTCOMES:
Change in Acceptance and Action Questionnaire (AAQ-II) | Change from Baseline psychological inflexibilty at 4 months
  'Acceptance and Action Questionnaire' assesses psychological inflexibility. It is a 7-item, seven-point Likert-type scale. Scores range between 7 and 49. Higher scores indicate higher levels of psychological inflexibility and worse outcome.
Change in Cognitive Fusion Questionnaire (CFQ) | Change from Baseline psychological inflexibilty at 4 months
  'Cognitive Fusion Questionnaire' assesses cognitive fusion (the tendency to believe the literal content of private events). It is a 7-item, seven-point Likert-type scale. Scores range between 7 and 49. Higher scores in the questionnaire indicate higher levels of cognitive fusion and worse outcome.
Change in Liebowitz Social Anxiety Scale LSAS | Change from Baseline psychological inflexibilty at 4 months
  'Liebowitz Social Anxiety Scale' assesses social anxiety. It is a 24-item, four-point Likert-type scale. Scores range between 0 and 72. Scores above 51 indicates significant social anxiety (González, Bascaran & Saiz, 2001). Higher the score in the questionnaire, indicate higher levels of social anxiety and worse outcome.
Change in Self-Statements during Public Speaking SSPS | Change from Baseline psychological inflexibilty at 4 months
  'Self-Statements during public Speaking questionnaire' assesses positive and negative self-statements. It is a 10-item, six-point Likert-type scale. It includes two subscales. Scores in positive self-statements subscale range between 5 and 30. Higher the score in this subscale, indicate higher levels of positive self-statements and better outcome. Scores in negative self-statements subscale range between 5 and 30. Higher the score in this subscale, indicate higher levels of negative self-statements and worse outcome.
Change in Public Speaking Self-efficacy and Fear Questionnaire CAHP | Change from Baseline psychological inflexibilty at 4 months
  'Public speaking self-efficacy and fear questionnaire' assesses public speaking self-efficacy and public speaking fear. It is a 12-item, six-point Likert-type scale. It includes two subscales (self-efficacy and fear). Scores in self-efficacy subscale range between 12 and 72. Higher the score in the sef-efficacy subscale, indicate higher levels of public speaking self-efficacy and better outcome. Scores in public speaking fear subscale range between 12 and 72. Higher the score in the fear subscale, indicate higher levels of public speaking fear and worse outcome.
Change in Anxiety intensity subjective scale | Change from Baseline psychological inflexibilty at 4 months
  'Anxiety intensity subjective scale' asesses global self-assessment of intensity of public speaking anxiety VAS-ratings (range from 0 = very low intensity to 10 = very high intensity). Higher the score in scale, indicate higher levels of public speaking anxiety intensity and worse outcome.
Change in Anxiety interference subjective scale | Through study completion, an average of 4 months
  'Anxiety interference subjective scale' assesses global self-assessment of interference of public speaking anxiety VAS-ratings (range from 0 = very low interference to 10 = very high interference). Higher the score in scale, indicate higher levels of public speaking anxiety interference and worse outcome.
Change in Change in Satisfaction with performance subjective scale | Through study completion, an average of 4 months
  'Satisfaction with performance subjective scale' assesses global self-assessment of satisfaction with performance VAS-ratings (range from 0 = very low satisfaction to 10 = very high satisfaction). Higher the score in scale, indicate higher satisfaction and better outcome.
Change in Behavioral Checklist for Performance Anxiety (Paul, 1966, adapted by Bados, 1986) | Through study completion, an average of 4 months
  Behavioral Checklist for Performance Anxiety assesses anxiety performance. It includes using video recordings, 'CODIMG' behavioral observation and analysis coding software. It is a 14-items checklist. Scores range between 0 and 14. Higher the score in the checklist, indicate higher levels of anxiety performance and worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Montesinos, Ph.D., Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT05573620/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT05573620/ICF_001.pdf